CLINICAL TRIAL: NCT00210106
Title: Treatment of Unresectable Colorectal Metastases by Radiofrequency Ablation Combined or Not With Resection, With or Without Neoadjuvant Chemotherapy. A Phase 2 Study.
Brief Title: Treatment of Unresectable Colorectal Metastases by Radiofrequency Ablation Combined or Not With Resection, With or Without Neoadjuvant Chemotherapy.
Acronym: ARF2003
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IB2003-11; ARF2003
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Results first posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-04

CONDITIONS: Colorectal Cancer
Keywords: Radiofrequency ablation; Colorectal cancer; Liver metastases
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intraoperative radiofrequency ablation (IRFA) (Experimental): IRFA treatment, either with or without resection, was performed at laparotomy within 28 days of inclusion in the study. The type of IRFA current generator and probes, and whether or not resection was performed, was at the discretion of the surgeon.
  Interventions: Device: Ablathermy

INTERVENTIONS:
Device: Ablathermy

SUMMARY:
The hypothesis is that radiofrequency ablation combined or not with resection may allow a local control (the liver) in patients suffering from unresectable colorectal liver metastases. Patients may have benefit or not from a preoperative (neoadjuvant) chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

Colorectal cancer Hepatic metastases unresectable by classical surgery Performance status < 2

Exclusion Criteria:

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2003-06; Primary Completion 2008-12 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Serge EVRARD, Pr, Principal Investigator — Institut Bergonié
Locations (12):
- France (12):
  - CHU d'Angers, Angers
  - Centre Saint Michel, Angoulême
  - CHU de Bordeaux, Bordeaux
  - Institut Bergonié - Centre Régional de Luttre Contre le Cancer de Bordeaux et du Sud Ouest, Bordeaux
  - Hopital Béclère, Clamart
  - Hopital Sub-Urbain du Bouscat, Le Bouscat
  - Hopital de la Croix Rousse, Lyon
  - Hopital Saint Eloi, Montpellier
  - Centre Hospitalier, Niort
  - Centre de Radiothérapie et d'Oncologie Médicale, Pau
  - Clinique Mutualiste de Pessac, Pessac
  - Clinique Francheville, Périgueux

REFERENCES:
- [Result] Evrard S, Rivoire M, Arnaud J-, Lermite E, Bellera C, Fonck M, Becouarn Y, Lalet C, Puildo M, Mathoulin-Pelissier S. Unresectable colorectal cancer liver metastases treated by intraoperative radiofrequency ablation with or without resection. Br J Surg. 2012 Apr;99(4):558-65. doi: 10.1002/bjs.8724. No abstract available. PMID 22396054

RESULTS

PARTICIPANT FLOW:
Groups:
- Intraoperative Radiofrequency Ablation (IRFA): IRFA treatment, either with or without resection, was performed at laparotomy within 28 days of inclusion in the study. The type of IRFA current generator and probes, and whether or not resection was performed, was at the discretion of the surgeon.
  Ablathermy
Period: Overall Study
Arm/Group | Intraoperative Radiofrequency Ablation (IRFA)
Started | 52
Safety Population (safety population is defined as patients who received IRFA treatment with our without resection.) | 49
Completed (Patients eligible (without major protocol deviation) who received the treatment (IRFA +/- surgery) and for whom 2 scans (2 months and 3 months) were available.) | 38
Not Completed | 14
Not completed — Death | 1
Not completed — Protocol Violation | 13

BASELINE CHARACTERISTICS:
Arm/Group | Intraoperative Radiofrequency Ablation (IRFA)
Number analyzed (Participants) | 52
Age, Continuous [Median (Full Range); unit: years] | 60 [30 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 40
Region of Enrollment [Number; unit: participants]
  France | 52

OUTCOME MEASURES:

1. Primary Outcome: Complete Hepatic Response Rate at 3 Months
Description: Complete hepatic response (CHR) rate was defined as the absence of new hepatic lesions or contrast enhancement at the ablation and resection sites on CT performed at 2 and 3 months. CHR at 3 months was reported
Time Frame: 3 months
Population: Patients evaluable for efficacy (completed) : eligible, treated and with 2 scans available
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Intraoperative Radiofrequency Ablation (IRFA)
Number analyzed (Participants) | 38
percentage of participants | 79 [63 to 90]

2. Secondary Outcome: Overall Survival
Description: OS was defined as the time from the treatment initiation to death due to any cause. Participants without documented death were censored at the date of the last follow-up or last patient contact. The OS was calculated using the product-limit (Kaplan-Meier) method for censored data. 1-year and 2-year OS rate were reported.
Time Frame: at 1 and 2 years
Population: Patients evaluable for efficacy (completed) : eligible, treated and with 2 scans available
Measure: Number (95% Confidence Interval); unit: percent probability of survival
Arm/Group | Intraoperative Radiofrequency Ablation (IRFA)
Number analyzed (Participants) | 38
percent probability of survival
  OS rate at 1 year | 97.4 [82.7 to 99.6]
  OS rate at 2 years | 91.7 [76.3 to 97.2]

3. Secondary Outcome: Event-free Survival
Description: Event-free survival was measured from the date of intervention to the date of the first of the following events: initial failure, disease progression (hepatic or distant) or death (all causes). Patients who were alive and event-free were consored at the last documented date of follow-up. 1-year and 2-years EFS rates were reported.
Time Frame: at 1 and 2 years
Population: Patients evaluable for efficacy (completed) : eligible, treated and with 2 scans available
Measure: Number (95% Confidence Interval); unit: percent probability of survival
Arm/Group | Intraoperative Radiofrequency Ablation (IRFA)
Number analyzed (Participants) | 38
percent probability of survival
  EFS rate at 1 year | 18.4 [8.1 to 32.0]
  EFS rate at 2 years | 10.5 [3.3 to 22.5]

ADVERSE EVENTS:
Time Frame: Adverse events were collected/monitored within 30 days after treatment and within 3 months post-treatment and deaths were monitored/assessed for up to 2 years post-treatment for each participant (in the scope of survival assessment)
Description: All adverse events observed in study participants were defined by the Clavien-Dindo classification system of surgical complications.
Arm/Group | Intraoperative Radiofrequency Ablation (IRFA)
All-Cause Mortality (participants affected / at risk) | 16/49
Serious Adverse Events (participants affected / at risk) | 5/49
Other Adverse Events (participants affected / at risk) | 6/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intraoperative Radiofrequency Ablation (IRFA) (N=49)
Thromboembolic event (Vascular disorders) | 1 (1)
Hepatic infection (Infections and infestations) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intraoperative Radiofrequency Ablation (IRFA) (N=49)
Duodenal obstruction (Gastrointestinal disorders) | 3 (3)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes